CLINICAL TRIAL: NCT03140137
Title: Retrospective Observational Study on the Safety of Immune Checkpoint Inhibitors in the Treatment of Advanced Melanoma and Lung Cancers in Patients With Pre-Existing Autoimmune Diseases
Brief Title: Immune Checkpoint Inhibitors and Pre-existing Autoimmune Diseases
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: CHECKAUTO
Record Dates: First submitted 2017-02-24; First posted 2017-05-04 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Autoimmune Diseases; Advanced Cancer
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Checkpoint inhibitor therapy — Treatment by ipilimumab, nivolumab or pembrolizumab for advanced cancer in clinical practice

SUMMARY:
The tolerance of immune checkpoint inhibitors is unknown in patients with pre-existing autoimmune conditions. This retrospective nation-wide study will assess their tolerance in patients with pre-existing autoimmune conditions who received immune checkpoint inhibitors for an advanced cancer in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Pre-existing autoimmune disease as diagnosed by the physician
* Immune checkpoint inhibitor therapy for an advanced cancer

Exclusion Criteria:

* Auto-immune disease developed only after the start of the immune checkpoint inhibitor therapy
* Absence of follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a pre-existing autoimmune disease who received immune checkpoint inhibitors for the treatment of an advanced cancer in clinical practice.
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2017-01-21 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2018-01-04 (Actual)

PRIMARY OUTCOMES:
Autoimmune disease flare | through study completion, an average of 1 year
  Increase in the activity of the pre-existing autoimmune disease as assessed by the treating physician

SECONDARY OUTCOMES:
Other immune/inflammatory complications | through study completion, an average of 1 year
  Development of a new immune/inflammatory condition after the start of the therapy

CONTACTS AND LOCATIONS:
Overall Officials: Divi CORNEC, Study Director — CHRU de Brest
Locations (5):
- France (5):
  - CH d'AIX, Aix-en-Provence
  - CHU de DIJON, Dijon
  - CHD Vendée, La Roche-sur-Yon
  - Ch Le Mans, Le Mans
  - CH de MACON, Mâcon